CLINICAL TRIAL: NCT06103188
Title: Comparing Melatonin to Diazepam as a Premedication: a Triple-blind, Randomized, Placebo Controlled Clinical Trial
Brief Title: Comparing the Effect of Melatonin, Diazepam, and Placebo on Decreasing the Level of Anxiety Preoperatively
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Omar Ismail, Principle Investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M001
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Anxiety; Preoperative Anxiety
Keywords: Preoperative anxiety; Anxiolytic; Melatonin; Diazepam; Sedation; Premedication
MeSH Terms: conditions — Anxiety Disorders | interventions — Diazepam; Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): A 5mg vitamin B12 pill
  Interventions: Drug: Placebo
- Diazepam (Active Comparator): A 5mg diazepam pill
  Interventions: Drug: Diazepam
- Melatonin (Experimental): A 5mg melatonin pill
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Placebo — The placebo pill will be given to the patients 1 hour prior to their planned surgery.
  Arms: Placebo
Drug: Diazepam — Diazepam will be given to the patients 1 hour prior to their planned surgery.
  Arms: Diazepam
Drug: Melatonin — Melatonin will be given to the patients 1 hour prior to their planned surgery.
  Arms: Melatonin

SUMMARY:
The goal of this clinical trial is to compare the effect of melatonin, diazepam, and placebo on the level of anxiety in patients undergoing surgery. The main question it aims to answer is:

• Is melatonin effective in reducing the anxiety of patients undergoing surgery? Participants will be asked to answer a questionnaire then they will receive either melatonin, diazepam, or placebo, and then after an hour, they will answer the same questionnaire again.

Researchers will compare melatonin, diazepam, and placebo to see if melatonin is as effective in reducing the level of anxiety as diazepam in patients undergoing surgery.

DETAILED DESCRIPTION:
Anxiety is a tense unpleasant sensation experienced by many individuals secondary to their concerns or due to the anticipation of an unpleasant experience like a surgery. Even with the advancement of medical treatment, preoperative anxiety remains a widespread complaint that affects the patients psychologically and physically, and at the same time adversely affecting the outcome of the operation and the experience of the patient.

In this triple-blind, randomized clinical study, we aim to compare melatonin to diazepam regarding its efficacy in reducing preoperative anxiety, as well as assessing multiple other effects such as sedation, orientation, and cognition, by applying validated tools to patients undergoing elective surgeries before and after administering the premedication.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2
* Posted for general anesthesia
* Aging between 18 and 65 years

Exclusion Criteria:

* Allergy to any of the drugs under study
* Pregnancy
* Illiteracy
* Any mental illness
* Taking antipsychotics, antidepressants, anxiolytics, or sedatives

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Ismail, Principal Investigator — University of Jordan
Locations (1):
- Jordan University Hospital, Amman, Jordan

REFERENCES:
- [Derived] Ismail O, Albdour K, Jaber K, Jaber Y, Alsaras A, Younis A, Froukh U, Momani Y, Abu-Halaweh S. The efficacy of melatonin as a preoperative anxiolytic in real-world setting: a randomized controlled trial. Hosp Pract (1995). 2025 Feb;53(1):2600245. doi: 10.1080/21548331.2025.2600245. Epub 2025 Dec 9. PMID 41346130

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Melatonin | Diazepam | Placebo
Started | 29 | 29 | 29
Completed | 28 | 23 | 25
Not Completed | 1 | 6 | 4
Not completed — Lost to Follow-up | 1 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin | Diazepam | Placebo | Total
Number analyzed (Participants) | 28 | 23 | 25 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 23 | 25 | 76
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [25 to 37] | 43 [33.5 to 52.5] | 37 [30 to 44] | 38.5 [29.5 to 47.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 10 | 39
  Male | 12 | 10 | 15 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 23 | 25 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Amsterdam Preoperative Anxiety and Information Scale [Median (Inter-Quartile Range); unit: units on a scale] — The Amsterdam Preoperative Anxiety and Information Scale consists of 6 items with the responses to each item ranging from a score of 1 to 5.
  The minimum score possible is 6 and the maximum score is 30, the higher the score the higher the anxiety level.
  The scale is the sum of two subscales:
  1. Need for Information subscale: consists of two items (minimum score of 2 and maximum score of 10, the higher the score the more need for information).
  2. Anxiety subscale: consists of four items (minimum score of 4 and maximum score of 20, the higher the score the higher the anxiety level).
  units on a scale
    Baseline APAIS | 10 [4 to 16] | 11 [7 to 15] | 6 [2 to 10] | 10 [4.5 to 15.5]
    Baseline APAIS Need for Information subscale | 3.5 [1.25 to 4.75] | 5 [3 to 7] | 2 [0 to 4] | 4 [1.75 to 6.25]
    Baseline APAIS Anxiety subscale | 7.5 [4.25 to 10.75] | 6 [4 to 8] | 4 [1.5 to 6.5] | 6 [3 to 9]
Baseline Visual Analogue Scale for Anxiety score (VAS-A) [Median (Inter-Quartile Range); unit: units on a scale] — VAS (Visual Analogue Score) Anxiety Scale is a 100 mm long scale. The scale is marked in millimeters from 0 to 100, where 0 correlates with no anxiety at all, and 100 correlates to anxiety as bad as possible. The maximum score is 100 and minimum 0. The patient is asked to point on the scale according to his anxiety level. The more the reduction in anxiety from baseline, the better the outcome.
  units on a scale | 10 [8 to 12] | 30 [12.5 to 47.5] | 20 [0 to 70] | 30 [10 to 50]
Baseline Ramsay sedation score [Median (Inter-Quartile Range); unit: units on a scale] — Ramsay sedation scale (RSS) is scored based on the level of sedation.
  It consists of six levels scored from 1 to 6:
  1. Patient is anxious and agitated or restless, or both
  2. Patient is cooperative, oriented, and tranquil
  3. Patient responds to commands only
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus
  6. Patient exhibits no response. As the patient becomes more sedated he receives a higher score on the scale (minimum of 1 and maximum of 6).
  units on a scale | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
Baseline orientation score [Median (Inter-Quartile Range); unit: units on a scale] — Orientation is assessed with a three-point scale as follows:
  0 - None
  1. - Orientation to either time or place
  2. - Orientation to both The higher the score the better the level of orientation. (minimum 0 and maximum of 2).
  units on a scale | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Change in the Anxiety Score Using the Visual Analogue Score for Anxiety Between Treatment Arms
Description: VAS (Visual Analogue Score) Anxiety Scale is a 100 mm long scale. The scale is marked in millimeters from 0 to 100, where 0 correlates with no anxiety at all, and 100 correlates to anxiety as bad as possible. The maximum score is 100 and minimum 0. The patient is asked to point on the scale according to his anxiety level. The more the reduction in anxiety from baseline, the better the outcome.
Time Frame: Before administration of premedication, and after 1 hour from the administration of the premedication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Melatonin | Diazepam | Placebo
Number analyzed (Participants) | 28 | 23 | 25
score on a scale | 0 [-5 to 5] | 0 [-5 to 5] | 0 [-7.5 to 7.5]

2. Primary Outcome: Change in Anxiety Score Based on The Amsterdam Preoperative Anxiety and Information Scale (APAIS) Between Treatment Arms
Description: The Amsterdam Preoperative Anxiety and Information Scale (APAIS) is a self-reported questionnaire. The scale consists of six items, four of which assess the patient's anxiety, while the last two assess the patients' need-for-information and the patient must choose how much he agrees with each item on a scale of 1 (not at all) to 5 (very much). The scores of each item are summed to provide the total score.
  The minimum score possible is 6 and the maximum score is 30, the higher the score the higher the anxiety level and need for information.
  The scale consists of two subscales:
  Need for Information subscale: consists of two items (minimum score of 2 and maximum score of 10, the higher the score the more need for information).
  Anxiety subscale: consists of four items (minimum score of 4 and maximum score of 20, the higher the score the higher the anxiety level).
  The total scale is the sum of the two subscales.
Time Frame: Before administration of premedication, and after 1 hour from the administration of the premedication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Melatonin | Diazepam | Placebo
Number analyzed (Participants) | 28 | 23 | 25
score on a scale
  APAIS difference | -0.5 [-2 to 1] | -1 [-3 to 1] | 0 [-1 to 1]
  Need for information subscale difference | 0 [-0.5 to 0.5] | 0 [-1.5 to 1.5] | 0 [-1 to 1]
  Anxiety subscale difference | 0 [-1.5 to 1.5] | 0 [-1 to 1] | 0 [-0.5 to 0.5]

3. Secondary Outcome: Change in Sedation Between Treatment Arms
Description: Ramsay sedation scale (RSS) is scored based on the level of sedation.
  It consists of six levels scored from 1 to 6:
  1. - Patient is anxious and agitated or restless, or both
  2. - Patient is cooperative, oriented, and tranquil
  3. - Patient responds to commands only
  4. - Patient exhibits brisk response to light glabellar tap or loud auditory stimulus
  5. - Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus
  6. - Patient exhibits no response.
  As the patient becomes more sedated he receives a higher score on the scale (minimum of 1 and maximum of 6).
Time Frame: Before administration of premedication, and after 1 hour from the administration of the premedication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Melatonin | Diazepam | Placebo
Number analyzed (Participants) | 28 | 23 | 25
score on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Change in Orientation Between Treatment Arms
Description: Orientation will be assessed with a three-point scale as follows:
  0 - None
  1. - Orientation in either time or place
  2. - Orientation in both
Time Frame: Before administration of premedication, and after 1 hour from the administration of the premedication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Melatonin | Diazepam | Placebo
Number analyzed (Participants) | 28 | 23 | 25
score on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

5. Other Pre Specified Outcome: Change in the Anxiety Score Using the Visual Analogue Score for Anxiety Between Genders
Description: as for outcome 1
Time Frame: Before administration of premedication, and after 1 hour from the administration of the premedication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Males: Only the male participants of the entire sample
- Females: Only the female participants of the entire sample.
Arm/Group | Males | Females
Number analyzed (Participants) | 37 | 39
score on a scale | 0 [0 to 0] | 0 [-10 to 10]

6. Other Pre Specified Outcome: Change in Anxiety Score Based on The Amsterdam Preoperative Anxiety and Information Scale (APAIS) Between Genders
Description: as for outcome 2
Time Frame: Before administration of premedication, and after 1 hour from the administration of the premedication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Males | Females
Number analyzed (Participants) | 37 | 39
score on a scale
  Difference on the APAIS scale | 0 [-1 to 1] | -1 [-3 to 1]
  Difference on the APAIS Need for Information subscale | 0 [0 to 0] | 0 [-1 to 1]
  Difference on the APAIS Anxiety subscale | 0 [0 to 0] | 0 [-1.5 to 1.5]

7. Other Pre Specified Outcome: Change in Sedation Between Genders
Description: Ramsay sedation scale (RSS) is scored based on the level of sedation.
  It consists of six levels scored from 1 to 6:
  1. Patient is anxious and agitated or restless, or both
  2. Patient is cooperative, oriented, and tranquil
  3. Patient responds to commands only
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus
  6. Patient exhibits no response.
  As the patient becomes more sedated he receives a higher score on the scale (minimum of 1 and maximum of 6).
Time Frame: Before administration of premedication, and after 1 hour from the administration of the premedication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Males | Females
Number analyzed (Participants) | 37 | 39
score on a scale | 0 [0 to 0] | 0 [0 to 0]

8. Other Pre Specified Outcome: Change in Orientation Between Genders
Description: as for outcome 4
Time Frame: Before administration of premedication, and after 1 hour from the administration of the premedication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Males | Females
Number analyzed (Participants) | 37 | 39
score on a scale | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Within one day of admission of the drug (until the participants were discharged home).
Arm/Group | Melatonin | Diazepam | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 0/28 | 0/23 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT06103188/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT06103188/SAP_001.pdf